CLINICAL TRIAL: NCT05007639
Title: A Public Health Intervention Program to Improve the Initial Management of Soft Tissue Sarcomas.
Acronym: IPSSAR
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB2008-IPSSAR
Record Dates: First submitted 2021-08-02; First posted 2021-08-16 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-11

CONDITIONS: Sarcoma
Keywords: publich health intervention programme
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients diagnosed BEFORE implementation of the public health intervention program: All adult patients (≥18 years old) diagnosed between 1 November 2006 and 31 December 2007 in the Aquitaine and Midi-Pyrénées administrative districts in South-West France (6 million inhabitants, 10% of the French population) with primary STS of any stage were included. Patients with visceral, bone, uterus or Kaposi's sarcoma, gastrointestinal stromal tumors, or mesotheliomas were not included. Patients being treated for recurrence, and patients diagnosed outside of the administrative districts were not eligible. STS diagnoses were made in public or private pathology laboratories. Data were collected from all relevant sources: pathology reports, medical records from private and public centers,
  Interventions: Other: No public Health intervention programme
- Patients diagnosed DURING implementation of the public health intervention program: Same eligibility criteria as for the group "before implementation of the public health intervention program", except that patients were diagnosed between 1 january 2008 and 31 october 2008.
- Patients diagnosed AFTER implementation of the public health intervention program: Same eligibility criteria as for the group "before implementation of the public health intervention program", except that patients were diagnosed between 1 November 2008 and 31 December 2009.
  Interventions: Other: Public Health intervention programme

INTERVENTIONS:
Other: Public Health intervention programme — The public health intervention programme combined 3 actions : a simple dissemination of information via the regional Unions of private practice physicians and the local correspondents of the regional networks (action 1), an action in the form of oral communication during regional meetings of professionals (action 2) and an action focused on each surgeon for whom the pathologist has diagnosed soft tissue sarcoma (action 3).
  Groups: Patients diagnosed AFTER implementation of the public health intervention program
Other: No public Health intervention programme
  Groups: Patients diagnosed BEFORE implementation of the public health intervention program

SUMMARY:
Sarcomas are rare tumours that represent less than 1% of cancers. Their actual incidence in France, however, is not known. The chances of survival at 5 years, without signs of the disease, are currently estimated at about 60%. The possibility of soft tissue sarcoma (STS) is frequently unrecognised, leading to an inappropriate initial diagnostic process and often to inadequate surgery. Compliance with good practice guides, which we can recall were targeted at oncologists, is good when the patient's record is discussed within the framework of a multidisciplinary consultation. The consequences of inadequate initial management, however, can be critical: unplanned surgery results in the need for systematic repeat procedure, with residual tumour found in more than half of cases, and the absence of multidisciplinary care has a deleterious impact on local disease control and specific survival.

The objective of the study is to measure the impact of a public health intervention programme focused on the initial management of STS among all professionals who may come to suspect or diagnose soft tissue sarcoma. For this project, the 4 regions involved in the Cancéropôle du Grand Sud-Ouest, France (Aquitaine, Languedoc-Roussillon, Limousin and Midi-Pyrénées) propose to implement actions targeted at general practitioners, treating physicians and non-specialist surgeons in the field of STS, aimed at improving initial care.

An improvement in initial management (diagnosis and assessment) which should allow an improvement in the loco-regional control of these diseases and in the specific survival of the patients. The actions recognised as effective in this study could then be adapted and extended to the rest of France via the French sarcomas group and the bone tumours study group (GSF-GETO).

DETAILED DESCRIPTION:
Background: Sarcomas are rare tumours that represent less than 1% of cancers. Their actual incidence in France, however, is not known. The chances of survival at 5 years, without signs of the disease, are currently estimated at about 60%. The possibility of soft tissue sarcoma (STS) is frequently unrecognised, leading to an inappropriate initial diagnostic process and often to inadequate surgery. Compliance with good practice guides, which we can recall were targeted at oncologists, is good when the patient's record is discussed within the framework of a multidisciplinary consultation. The consequences of inadequate initial management, however, can be critical: unplanned surgery results in the need for systematic repeat procedure, with residual tumour found in more than half of cases, and the absence of multidisciplinary care has a deleterious impact on local disease control and specific survival.

Objectives: The objective of the study is to measure the impact of a public health intervention programme focused on the initial management of STS among all professionals who may come to suspect or diagnose soft tissue sarcoma. For this project, the 4 regions involved in the Cancéropôle du Grand Sud-Ouest, France (Aquitaine, Languedoc-Roussillon, Limousin and Midi-Pyrénées) propose to implement actions targeted at general practitioners, treating physicians and non-specialist surgeons in the field of STS, aimed at improving initial care.

Outline: This is a "before and after (the intervention programme)" study with a "control" group (Nantes region with multidisciplinary "sarcoma" consultation meetings organised, but where no specific intervention shall be made).

Course the intervention: The programme shall combine 3 actions: a simple dissemination of information via the regional Unions of private practice physicians and the local correspondents of the regional networks (action 1), an action in the form of oral communication during regional meetings of professionals (action 2) and an action focused on each surgeon for whom the pathologist has diagnosed soft tissue sarcoma (action 3).

Study size: It is assumed that the proposed programme shall serve to measure a 35% improvement in the proportion of adequate care (70% with intervention versus 35%). To take into account in the analysis of potential clusters of practices (professionals with similar medical practices), the number of subjects was increased to 60 observations per study phase (before/after). The results of the "Before the intervention" study should enable us to adjust the number of subjects to take into account any cluster effects, which cannot be estimated as it is, while taking into account the feasibility since these are rare tumours.

Endpoints: For each patient, the main analyses shall focus on different care quality endpoints, in particular those relating to the initial diagnosis and initial surgery stages. The elements of these endpoints shall be collected in health establishments and pathology laboratories in the regions involved.

Impacts and perspectives: An improvement in initial management (diagnosis and assessment) which should allow an improvement in the loco-regional control of these diseases and in the specific survival of the patients. The actions recognised as effective in this study could then be adapted and extended to the rest of France via the French sarcomas group and the bone tumours study group (GSF-GETO).

ELIGIBILITY:
Inclusion Criteria:

* Primary soft-tissue sarcoma (STS)
* any stage

Exclusion Criteria:

* Patients with visceral, bone, uterus or Kaposi's sarcoma, gastrointestinal stromal tumors, or mesotheliomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥18 years old) diagnosed between 1 November 2006 and 31 December 2009 in the Aquitaine and Midi-Pyrénées administrative districts in South-West France (6 million inhabitants, 10% of the French population) with primary STS of any stage were included.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2006-11-02 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simone MATHOULIN-PELISSIER, MD, PhD, Principal Investigator — Institut Bergonié, COmprehensive Cancer Center, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mathoulin-Pelissier S, Chevreau C, Bellera C, Bauvin E, Saves M, Grosclaude P, Albert S, Goddard J, Le Guellec S, Delannes M, Bui BN, Mendiboure J, Stoeckle E, Coindre JM, Kantor G, Kind M, Cowppli-Bony A, Hoppe S, Italiano A. Adherence to consensus-based diagnosis and treatment guidelines in adult soft-tissue sarcoma patients: a French prospective population-based study. Ann Oncol. 2014 Jan;25(1):225-31. doi: 10.1093/annonc/mdt407. Epub 2013 Nov 26. PMID 24285018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All adult patients (≥18 years old) diagnosed between 1 November 2006 and 31 December 2007 in the Aquitaine and Midi-Pyrénées administrative districts in South-West France (6 million inhabitants, 10% of the French population) with primary STS of any stage were included.
Groups:
- Patients Diagnosed BEFORE Implementation of the Public Health Intervention Program: All adult patients (≥18 years old) diagnosed between 1 November 2006 and 31 December 2007 in the Aquitaine and Midi-Pyrénées administrative districts in South-West France (6 million inhabitants, 10% of the French population) with primary STS of any stage were included. Patients with visceral, bone, uterus or Kaposi's sarcoma, gastrointestinal stromal tumors, or mesotheliomas were not included. Patients being treated for recurrence, and patients diagnosed outside of the administrative districts were not eligible. STS diagnoses were made in public or private pathology laboratories. Data were collected from all relevant sources: pathology reports, medical records from private and public centers,
  Public Health intervention programme: The public health intervention programme combined 3 actions : a simple dissemination of information via the regional Unions of private practice physicians and the local correspondents of the regional networks (action 1), an action in the form of oral communication during regional meetings of professionals (action 2) and an action focused on each surgeon for whom the pathologist has diagnosed soft tissue sarcoma (action 3).
  No public Health intervention programme
Period: Overall Study
Arm/Group | Patients Diagnosed BEFORE Implementation of the Public Health Intervention Program
Started | 274
Completed | 274
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Diagnosed BEFORE Implementation of the Public Health Intervention Program
Number analyzed (Participants) | 274
Age, Continuous [Median (Full Range); unit: years] | 63.8 [18 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 158
Region of Enrollment [Count of Participants; unit: Participants]
  France | 274

OUTCOME MEASURES:

1. Primary Outcome: Adherence Rate to Diagnosis Imaging Guidelines for Patients With a Deep Sarcoma Tumor (Before Implementation of the Public Health Intervention Programme.
Description: Imaging criterion for patients with a deep tumor was considered "compliant" if patients received magnetic resonance imaging (MRI) or scan of the tumor zone before surgery.
  Adherence rate was calculated as the number of patients with "compliant imaging criterion" among patients with a deep tumor.
Time Frame: Assessed at surgery
Population: Participants analyzed : patients with a deep tumor
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Diagnosed BEFORE Implementation of the Public Health Intervention Program
Number analyzed (Participants) | 178
Participants | 145

2. Primary Outcome: Adherence Rate to Diagnosis Imaging Guidelines for Patients With a Superficial Sarcoma Tumor (Before Implementation of the Public Health Intervention Programme)
Description: Imaging criterion for patients with a superficial tumor was considered "compliant" if patients received an MRI, scan, or ultrasound before surgery.
  Adherence rate was calculated as the number of patients with "compliant imaging criterion" among patients with a superficial tumor.
Time Frame: Assessed at surgery
Population: Participants Analyzed: patients with a superficial tumor
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Diagnosed BEFORE Implementation of the Public Health Intervention Program
Number analyzed (Participants) | 89
Participants | 33

3. Primary Outcome: Adherence Rate to Diagnosis Technique (Biopsy) Guidelines for Patients With Deep Tumors Over 5 cm in Size or Tumors <5 cm Increasing in Size (Before Implementation of the Public Health Intervention Programme)
Description: Diagnosis technique (biopsy) was considered "compliant" for deep tumors over 5 cm in size or tumors <5 cm increasing in size if the diagnosis was made from a percutaneous or surgical biopsy.
  Adherence rate was calculated as the number of patients with "compliant diagnosis technique" among patients with deep tumors over 5 cm in size or tumors <5 cm increasing in size.
Time Frame: Assessed up to 2 months following diagnosis
Population: Participants Analyzed: patients with a deep tumor over 5 cm in size or tumors <5 cm increasing in size
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Diagnosed BEFORE Implementation of the Public Health Intervention Program
Number analyzed (Participants) | 232
Participants | 120

4. Primary Outcome: Adherence Rate to Discussion in Multidisciplinary Team Meeting (Before Implementation of the Public Health Intervention Programme)
Description: Discussion in multidisciplinary team (MDT) meeting was considered "compliant" if the patient record was discussed in MTD meeting before biopsy.
  Adherence rate was calculated as the number of patients with "compliant MDT meeting" among sarcoma patients with a biopsy.
Time Frame: Assessed up to 2 months prior to biopsy
Population: Participants Analyzed: patients with a biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Diagnosed BEFORE Implementation of the Public Health Intervention Program
Number analyzed (Participants) | 157
Participants | 10

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Patients Diagnosed BEFORE Implementation of the Public Health Intervention Program
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes